CLINICAL TRIAL: NCT00672581
Title: An Open-label Comparative Study of the Pharmacokinetics, Safety and Tolerability of ZD4054 (Zibotentan) Following a 10 mg Single Oral Dose of ZD4054(Zibotentan) to Healthy Subjects and to Subjects With Mild, Moderate and Severe Hepatic Impairment
Brief Title: Pharmacokinetics, Safety & Tolerability of ZD4054 (Zibotentan) in Subjects With Normal, Mild, Moderate and Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Thomas Morris, Medical Science Director, ZD4054, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4320C00025; 4054IL/0025
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment
MeSH Terms: interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Control (healthy volunteers)
  Interventions: Drug: ZD4054
- 2 (Experimental): Mild Hepatic Impairment
  Interventions: Drug: ZD4054
- 3 (Experimental): Moderate Hepatic Impairment
  Interventions: Drug: ZD4054
- 4 (Experimental): Severe Hepatic Impairment
  Interventions: Drug: ZD4054

INTERVENTIONS:
Drug: ZD4054 — 10mg, Oral tablet, single dose
  Other Names: Zibotentan

SUMMARY:
This study is designed to compare how ZD4054 (Zibotentan) is taken up, how it is broken down and removed from the body in subjects with liver cirrhosis and hepatic impairment compared to healthy subjects of a similar age, sex and weight. As for all clinical trials, safety and tolerability of the drug will be evaluated as well to develop dosing recommendations for dosing of ZD4054 (Zibotentan) in subjects with varying stages of hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Hepatically impaired subjects - Subjects with stable liver cirrhosis and hepatic impairment for at least 3 months prior to the start of the study.
* Healthy volunteers - Clinical laboratory tests within the normal reference range or results with minor deviations which are not considered by the Investigator to be clinically significant

Exclusion Criteria:

* In the opinion of the investigator, any evidence of additional severe or uncontrolled systemic disease (eg, cardiac, or renal disease) or evidence of any other significant clinical disorder or laboratory finding
* Healthy volunteers - History or presence of hepatic disease known to interfere with absorption, distribution, metabolism or excretion of drug
* Hepatically impaired subjects - Fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-04; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Characterise the pharmacokinetic profile of ZD4054 (Zibotentan) following a single 10 mg oral dose in subjects with normal hepatic function and in subjects with varying degrees of hepatic impairment. | predose and 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours post-dose

SECONDARY OUTCOMES:
Assess the safety of Zibotentan following a single 10 mg oral dose in subjects with normal hepatic function and in subjects with varying degrees of hepatic impairment by assessment of vital signs, ECG, clinical chemistry, haematology and adverse events. | Predose until post-study medical
Explore changes in protein binding of Zibotentan and the subsequent effects on its pharmacokinetics in subjects with normal hepatic function and in subjects with varying degrees of hepatic impairment by assessment of free Cmax, free AUC and unbound CL/F. | 3 hour post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Morris, Study Director — AstraZeneca, Medical Science Director; Blanka Cieslarova, MD, Principal Investigator — Medical Director & Head of Clinical Unit, PRA International
Locations (1):
- Research Site, Prague, Czechia

REFERENCES:
- [Derived] Tomkinson H, Kemp J, Oliver S, Swaisland H, Taboada M, Morris T. Pharmacokinetics and tolerability of zibotentan (ZD4054) in subjects with hepatic or renal impairment: two open-label comparative studies. BMC Clin Pharmacol. 2011 Mar 17;11:3. doi: 10.1186/1472-6904-11-3. PMID 21414193